CLINICAL TRIAL: NCT01775215
Title: A Comparative Study of Advanced Imaging Techniques in Predicting the Clinical Outcome in Aortic Stenosis
Brief Title: A Comparison of Advanced Imaging Techniques in Aortic Stenosis
Acronym: AIm-AS
Status: Withdrawn | Type: Observational
Why Stopped: Abandoned
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 12/LO/1846
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Aortic Stenosis
Keywords: Left Ventricular Function; Aortic Valve Replacement; Late Gadolinium Enhancement; Cardiac I123 MIBG; Longitudinal Strain; Brain Natriuretic Peptide; High Sensitivity Troponin I
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum sample.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A - Symptomatic severe AS: Patients with symptomatic severe aortic stenosis (AS) as per ESC guidelines, requiring aortic valve replacement.
  Interventions: Radiation: Cardiac I123-MIBG Scintigraphy; Other: Cardiac MRI; Other: Stress and rest Echocardiogram; Other: High Sensitivity Troponin I; Other: Brain Natriuretic Peptide
- B - Asymptomatic moderate to severe AS: Asymptomatic patients with moderate to severe aortic stenosis (AS) as per ESC guidelines ,with Left Ventricular ejection fraction >50%, not yet requiring aortic valve replacement.
  Interventions: Radiation: Cardiac I123-MIBG Scintigraphy; Other: Cardiac MRI; Other: Stress and rest Echocardiogram; Other: High Sensitivity Troponin I; Other: Brain Natriuretic Peptide

INTERVENTIONS:
Radiation: Cardiac I123-MIBG Scintigraphy
Other: Cardiac MRI
Other: Stress and rest Echocardiogram
Other: High Sensitivity Troponin I
Other: Brain Natriuretic Peptide

SUMMARY:
In patients with aortic stenosis the valve through which blood is pumped out of the main heart chamber is narrowed. This results in heart muscle working harder to open the valve so blood can circulate around the body. The muscle adapts to the increased pressure load to maintain efficiency. This can cause long-term muscle damage. To predict when this deterioration will require a valve replacement is difficult and untimely operation exposes patients to unnecessary risk.

We aim to compare all validated techniques looking at different aspects of heart muscle strain in these patients. These will be a blood sample measuring a specific hormone (BNP) and enzyme (Troponin), a nuclear scan to assess nerve activation, an MRI identifying scarring and an exercise echocardiogram that measures heart muscle response and pressure changes across the valve. Tests will be performed at recruitment and either after one year or after valve replacement, which ever comes first.

In comparing these different imaging techniques we aim to identify patients who will benefit from an early operation, those whose muscle is likely to recover back to normal and which patients it is safe to wait longer for the surgery, avoiding unnecessary risk.

The results of the study will benefit patients as it will help doctors more accurately assess the timing of valve surgery and improve their prediction of long term heart muscle recovery. It may also increase convenience in clinical management by reducing unnecessary tests and hospital trips. This would translate into cost savings for the NHS.

ELIGIBILITY:
Inclusion Criteria:

(Group A)

* Asymptomatic patients with moderate to severe Aortic Stenosis
* Ejection fraction greater than 50%
* Not yet being considered for valve surgery

(Group B)

* Severe Aortic Stenosis (as per ESC guidelines)
* Listed for immediate aortic valve replacement

Exclusion Criteria: (Group A and B)

* Inability to provide informed consent
* Concurrent primary valve lesions greater than mild (as defined by ESC criteria)
* Previous myocardial infarction (regional wall motion abnormality on resting echo)
* Cardiomyopathy
* Congenital heart disease
* Previous cardiac surgery
* Renal failure (CKD stage 3, eGFR >30ml/min/1.73m2)
* Pregnancy, risk of pregnancy, breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care Outpatient population under regular follow by either cardiology or cardio thoracic team.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Need for aortic valve replacement | 1 year

SECONDARY OUTCOMES:
Improvement in measured indices post aortic valve replacement | 6 months

OTHER OUTCOMES:
The change in rate of measured indices over time | 6 months - 1 year
The relative change in measured indices between each other over time | 6 months - 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kelion, MRCP DM, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (1):
- Harefield Hospital, London, United Kingdom